CLINICAL TRIAL: NCT02792205
Title: Performance Evaluation of Von Willebrand:Collagen-Binding Assays to Diagnose Von Willebrand Factor Deficiency in Patients With Increased Risk of Bleeding
Acronym: PERICOLL
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC16_0028
Record Dates: First submitted 2016-06-02; First posted 2016-06-07 (Estimated); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Von Willebrand Disease
Keywords: Willebrand factor deficiency; hematology; Willebrand:Collagen-binding
MeSH Terms: conditions — von Willebrand Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Non interventional study — no intervention

SUMMARY:
Von Willebrand Disease (VWD) is defined as an inherited bleeding disorder that is caused by deficiency or dysfunction of von Willebrand factor (VWF), a plasma protein that mediates the initial adhesion of platelets at sites of vascular injury and also binds and stabilizes blood clotting factor VIII (FVIII) in the circulation. The most severe forms of VWD are usually easy to diagnose (obvious hemorrhagic symptoms and major VWF deficiency), whereas the mild forms of the disease are still difficult to confirm. It is indeed reported that about 1% of the population carry mild biological VWF deficiency without any bleeding tendency and any "actual disease". On the contrary, some patients with severe bleeding history can carry a true VWF abnormality, well-confirmed by genetic studies, without any VWF deficiency when evaluated with standard biological methods, such as Ristocetin Cofactor activity (VWF:RCo). However, in these patients, the use of alternative methods, such as PFA-100 (Platelet Fonction Analyzer-100), the study of Factor VIII (FVIII:C) to VWF (FVIII:C/VWF) ratio or the evaluation of VWF activity using more specialized methods such as VWF:CB (VWF-Collagen Binding) assay can detect the VWF deficiency and possible hemorrhagic predisposition.

In this project, the investigators plan to assess the performance of VWF:CB in the diagnosis of VWF deficiency in patients with unexplained bleeding history.

ELIGIBILITY:
Inclusion Criteria:

* Patient with bleeding history sent to the Hemophilia Treatment Center in Dijon or Nantes University Hospital with abnormal bleeding score (>3 in men and >5 in women
* Patient who has provided a signed consent to participate at this study and for blood sampling
* Affiliation with French social security system

Non-Inclusion Criteria:

* Minors will not be included in the study.
* On-going pregnancy and postpartum period (3 months after delivery)
* Substitutive treatment with coagulation factor concentrates or desmopressin administration within 10 days before sampling.
* Ongoing infectious or inflammatory disease that can modify VWF levels.
* Diagnosis of obvious hemostasis disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study plans to enroll 200 patients (100 per Center) in a 2-year period. The recruitment will occur in standard consultation activity of the 2 Hemostasis Centers of Dijon and Nantes. As each Center carries out about 1200 consultations/year, this projection appears as feasible, since a majority of them are induced by hemorrhagic profile. Such a number of patients will allow reliable statistical analysis.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Von Willebrand factor levels measured with Von Willebrand factor: Collagen-Binding methods | Up to 1 year
  Deficiency is defined when VWF level is < 50IU/dL, as usually defined by Favaloro E.J. (2000).
  A composite reference standard (CRS) will be used to improve the imperfect Gold Standard (VWF: RCo). CRS will be defined as being positive if either VWF: RCo, VWF:Ag, PFA-100 or FVIII:C will be positive and negative otherwise.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Trossaërt, Dr, Principal Investigator — Nantes University Hospital
Locations (2):
- France (2):
  - Dijon University Hospital, Dijon
  - Nantes University Hospital, Nantes

IPD SHARING:
Plan to Share IPD: No